CLINICAL TRIAL: NCT03899428
Title: A Randomized, Open-label Trial Comparing Immune Checkpoint Therapy vs Target Therapy in Reducing Serum HBsAg Levels in Patients With HBeAg-positive Advanced Stage Hepatocellular Carcinoma (VICI-5)
Brief Title: Immune Checkpoint Therapy vs Target Therapy in Reducing Serum HBsAg Levels in Patients With HBsAg+ Advanced Stage HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Humanity & Health Medical Group Limited (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VICI-5
Record Dates: First submitted 2019-03-26; First posted 2019-04-02 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; Sorafenib; lenvatinib; regorafenib; cabozantinib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immune Checkpoint Therapy (Experimental): The subjects will receive durvalumab 1500 mg Q4W
  Interventions: Drug: Durvalumab
- Target Therapy (Experimental): The subjects will receive tyrosine kinase inhibitors, including sorafenib, lenvatinib, regorafenib, or cabozantinib, daily
  Interventions: Drug: Sorafenib; Drug: Lenvatinib; Drug: Regorafenib; Drug: Cabozantinib

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 mg IV (intravenous infusion)
  Other Names: IMFINZI®
  Arms: Immune Checkpoint Therapy
Drug: Sorafenib — Prescribed by physician.
  Other Names: Nexavar, BAY43-9006
  Arms: Target Therapy
Drug: Lenvatinib — Prescribed by physician.
  Other Names: Lenvima, E7080
  Arms: Target Therapy
Drug: Regorafenib — Prescribed by physician.
  Other Names: Stivarga, BAY73-4506
  Arms: Target Therapy
Drug: Cabozantinib — Prescribed by physician.
  Other Names: Cabometyx, XL184
  Arms: Target Therapy

SUMMARY:
It is estimated that over 50% of HCC cases worldwide are related to chronic HBV. There are approximately 350-400 million people across the world infected with HBV, the majority reside in or originate from Asia. Each year HBV accounts for 749,000 new cases of HCC and 692,000 HCC-related deaths. The annual incidence of HCC is estimated to be <1% for non-cirrhotic HBV infected patients and 2-3% for those with cirrhosis.

While the most approved nucleos(t)ide analogues (NA) suppress HBV replication through inhibition of HBV-DNA polymerase and are reported to reduce the risk of HCC incidence, however, such risk is not completely eliminated under NA treatment. The recent availability of commercial quantitative assays of serum hepatitis B surface antigen (HBsAg) has enabled quantitative HBsAg to be used as a biomarker for prognosis and treatment response in CHB. It has been suggested that HBsAg decline during lamivudine or entecavir therapy is slower and less pronounced compared to interferon treatment, despite a higher effect on HBV DNA suppression. Based on HBsAg kinetics, it has been estimated that the predicted median time to HBsAg loss in patients treated with lamivudine or entecavir is more than 30 years. Thus, treatment that can induce rapid decline of HBsAg would have clear advantage in reducing the treatment duration required to achieve HBsAg-loss.

Interestingly, in a recent preliminary study, 12-weeks of treatment with nivolumab has showed the modest effect on HBsAg decline in HBeAg negative CHB patients. Thus, in this clinical trial, the investigator will investigate whether immune checkpoint therapy is more effective in inducing HBsAg decline compared with target therapy in HBsAg-positive patients with advanced stage HCC.

ELIGIBILITY:
Inclusion Criteria:

1. HBsAg positive with serum HBsAg levels ≥ 2 log IU/ml
2. Age ≥ 18 years old on the day of consent
3. Capable of understanding and complying with the protocol requirements and signed informed consent
4. Documented histological or cytological diagnosis of HCC within 1 year
5. Barcelona Clinic Liver Cancer (BCLC) stage B (that is not eligible for locoregional therapy) or stage C
6. Child-Pugh Score class A or B
7. ECOG performance status of 0 or 1 at enrollment.
8. Treated with either entecavir or tenofovir or TAF before initiation of anti-PDL1 or TKI
9. At least 1 measurable lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have a short axis ≥15 mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), and that is suitable for accurate repeated measurements as per RECIST 1.1 guidelines. A lesion which progressed after previous ablation or TACE could be measurable if it meets these criteria
10. Adequate organ and marrow function, as defined below. Criteria "a," "b," "c," and "f" cannot be met with transfusions, infusions, or growth factor support administered within 14 days of starting the first dose.

    1. Hemoglobin ≥9 g/dL
    2. Absolute neutrophil count ≥1000/μL
    3. Platelet count ≥75000/μL
    4. Total bilirubin (TBL) ≤2.0× upper limit of normal (ULN)
    5. AST and ALT ≤5×ULN
    6. Albumin ≥2.8 g/dL
    7. International normalized ratio (INR) ≤1.6
    8. Calculated creatinine clearance ≥50 mL/minute as determined by Cockcroft-Gault (using actual body weight) or 24-hour urine creatinine clearance

Exclusion Criteria:

1. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
2. Radiation therapy within 4 weeks (2 weeks for radiation for bone metastases) or radionuclide treatment (eg, I-131 or Y-90) within 6 weeks of starting treatment. Subject is excluded if there are any clinically relevant ongoing complications from prior radiation therapy
3. Prior interferon treatment
4. Concomitant anticoagulation, at therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, low molecular weight heparin (LMWH), thrombin or coagulation factor X (FXa) inhibitors, or antiplatelet agents (eg, clopidogrel). Low-dose aspirin for cardioprotection (per local applicable guidelines), low-dose warfarin (≤ 1 mg/day), and low-dose LMWH are permitted.
5. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   a. Cardiovascular disorders including i. Symptomatic congestive heart failure, unstable angina pectoris, or serious cardiac arrhythmias ii. Uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic, or > 100 mm Hg diastolic despite optimal antihypertensive treatment iii. Stroke (including TIA), myocardial infarction, or other ischemic event within 6 months before starting treatment iv. Thromboembolic event within 3 months before starting treatment. Subjects with thromboses of portal/hepatic vasculature attributed to underlying liver disease and/or liver tumor are eligible b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: i. Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction ii. Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before starting treatment, Note: Complete healing of an intra-abdominal abscess must be confirmed prior to starting treatment c. Major surgery within 2 months before starting treatment. Complete healing from major surgery must have occurred 1 month before starting treatment. Complete healing from minor surgery (eg, simple excision, tooth extraction) must have occurred at least 7 days before starting treatment. Subjects with clinically relevant complications from prior surgery are not eligible d. Cavitating pulmonary lesion(s) or endobronchial disease e. Lesion invading a major blood vessel (eg, pulmonary artery or aorta) f. Clinically significant bleeding risk including the following within 3 months of starting treatment: hematuria, hematemesis, hemoptysis of >0.5 teaspoon (>2.5 mL) of red blood, or other signs indicative of pulmonary hemorrhage, or history of other significant bleeding if not due to reversible external factors g. Other clinically significant disorders such as: i. known infection with human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)-related illness requiring systemic treatment ii. Serious non-healing wound/ulcer/bone fracture iii. Malabsorption syndrome iv. Uncompensated/symptomatic hypothyroidism v. Requirement for hemodialysis or peritoneal dialysis
6. Subjects with untreated or incompletely treated varices with bleeding or high risk for bleeding are excluded with the following clarification: subjects with history of prior variceal bleeding must have been treated with adequate endoscopic therapy without any evidence of recurrent bleeding for at least 6 months prior to study entry and must be stable on optimal medical management (e.g. non-selective beta blocker, proton pump inhibitor) at study entry.
7. Moderate or severe ascites
8. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 7 days before starting treatment Note: If the QTcF is > 500 ms in first ECG, a total of 3 ECGs should be performed. If the average of these 3 consecutive results for QTcF is ≤ 500 ms, the subject meets eligibility in this regard.
9. Inability to swallow tablets
10. Previously identified allergy or hypersensitivity to components of the study treatment formulations
11. Pregnant or lactating females
12. Diagnosis of another malignancy within 2 years before starting treatment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to decline to ≥ 2 log10 IU/mL of serum HBsAg | Assessed up to 2 years

SECONDARY OUTCOMES:
Time to loss of serum HBsAg | Assessed up to 2 years
Time to development of anti-HBsAg | Assessed up to 2 years
Progression-free survival (PFS) per RECIST 1.1 | From date of starting treatment until the date of objective disease progression or death, assessed up to 2 years.
Objective response rate (ORR) per RECIST 1.1 | From date of starting treatment until the date of objective disease progression or death, assessed up to 2 years.
Overall survival (OS) | From the date of starting treatment until death due to any cause, assessed up to 2 years.
Adverse events assessed in terms of seriousness, severity, and relationship to the study material according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | From the time of signature of informed consent, throughout the treatment period, and up to the follow-up period, assessed up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, PhD, Principal Investigator — Humanity & Health Research Centre
Locations (1):
- Humanity & Health Research Centre, Hong Kong, Hong Kong SAR, Hong Kong

IPD SHARING:
Plan to Share IPD: No